CLINICAL TRIAL: NCT02153034
Title: A Study of the Pathogenesis and Management of M. Ulcerans Disease, Buruli Ulcer
Brief Title: Pathogenesis and Management of M. Ulcerans Disease, Buruli Ulcer
Acronym: Buruli_Path
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dr Richard Phillips, Dr, Kwame Nkrumah University of Science and Technology
Other Study IDs: MR/J01477X/1
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Buruli Ulcer; Mycobacterium Ulcerans Disease
Keywords: Buruli ulcer; Mycobacterium ulcerans disease; M. ulcerans disease
MeSH Terms: conditions — Buruli Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Buruli ulcer patients, no intervention: Buruli ulcer patients administered standard standard care by the attending physician
- Healthy contacts, no intervention: Healthy volunteers who will be contacts of patients recruited or non-endemic controls. No intervention will be administered

SUMMARY:
Buruli ulcer is a neglected tropical disease caused by infection with Mycobacterium ulcerans (Mu) in rural parts of West Africa. It causes large skin ulcers mainly in children aged 5 to 15 years. Access to treatment is limited and many cases present late. There have been major advances in understanding the mechanism of disease together with improved diagnosis and management. The aim of the proposed studies is to identify markers predictive of a rapid response to antibiotic treatment and to investigate the pathogenesis of paradoxical reactions and oedematous lesions in Mu disease.

Infection with Mu results in a nodule under the skin which enlarges and breaks down to form an ulcer. This is because Mu produces a toxin that spreads outwards and damages subcutaneous tissue. In recent years it has been found that antibiotic treatment for 8 weeks with daily tablets and intramuscular injections heals ulcers. This is unpleasant and it would be better if the treatment could be shortened. Our previous studies suggest this may be possible. Therefore a wide range of tests will be investigated in order to identify markers for people in whom the infection is at an early stage with low numbers of Mu bacteria and low levels of toxin in the skin. During antibiotic treatment the rate of healing will be measured to find out which markers are the most reliable.

In some patients new areas of inflammation develop despite treatment and this is called a paradoxical reaction. The immune response to Mu will be investigated serially during antibiotic treatment to investigate the cause of paradoxical reactions.

About 15% of patients have oedematous disease, the most severe form of Buruli ulcer. We will study the amount of Mu toxin produced by the strain of Mu cultured from patients with this form of the disease.

Hypothesis

* Buruli ulcer patients that heal rapidly/slowly or develop paradoxical reactions with treatment will have associated predictive viability or serum biomarkers.
* Buruli ulcer patients with oedematous disease are associated with larger amounts of mycolactone and viable organisms

DETAILED DESCRIPTION:
Procedures

Infected Participants

After collection of demographic data using standard World Health Organisation forms (BU01) together with a careful history to establish when early lesions (nodules, plaques and ulcers) were first observed, the type and dimensions of lesions will be documented together with digital photographs and tracings onto acetate sheets. For oedematous lesions only digital photographs will be obtained. Patients will be reviewed at 2 weekly intervals during standard antibiotic treatment (rifampicin 10mg/kg and streptomycin 15mg/kg) with further recordings of clinical data as is done for all routine patients. These measurements will enable calculation of rate of healing and healing time in relation to lesion size and type. Patients will be monitored for paradoxical reactions that occur after the start of treatment in about 8% of patients. These procedures are routinely provided as part of routine care of Buruli ulcer patients.

Samples

The additional samples required from patients for the study are an extra volume of blood (7ml) and 3 swabs taken on occasions (at baseline, week 4, 8, 12 and 16) only when the patient has a lesion at these time points. Swabs/fine needle aspirates are required to determine if organisms detected by polymerase chain reaction (PCR) are still viable, one for M. ulcerans culture, one for measurement of mycolactone concentration, and one for combined 16S ribosomal ribonucleic acid (rRNA) reverse transcriptase / insertion sequence IS2404 Real-Time qPCR assay (1).

For patients that develop paradoxical lesions during therapy an additional blood sample and 3 swabs/fine needle aspirates will be obtained at the time of the reaction for viability markers (M. ulcerans culture, combined 16S rRNA reverse transcriptase / IS2404 Real-Time quantitative polymerase chain reaction (qPCR) assay and mycolactone detection).

For oedematous lesions, one swab/fine needle aspirates will be obtained for mycolactone detection and quantification from lesions that are ulcerated. A 3 mm punch biopsy will be performed under local anaesthetic on non-ulcerated lesions for the same purpose only when the patient is 15 years old or above.

Established practice for routine diagnosis of M. ulcerans infection is to take fine needle aspirates from non-ulcerated lesions for acid-fast bacillus (AFB) detection, culture and PCR for IS2404. This specimen is not large enough for mycolactone quantification, an important part of the investigation into the pathogenesis of oedematous disease which often presents without ulceration. Swabs are used in the diagnosis of ulcers.

Controls For the household contacts of patients in endemic villages and healthy controls in non-endemic villages a 7ml blood sample will be obtained to investigate protein biomarkers by Luminex assay, T cell subsets by flow cytometry and immune responses using Enzyme Linked Immunosorbent Assay(ELISA) in a whole blood assay for comparative studies. No tissue biopsies will be taken.

Definition of paradoxical reaction Paradoxical reaction will be defined as an increase in inflammatory changes with increase in lesion size of greater than 100%, after initial improvement and decrease in size; and/or the appearance of new lesions following or during antimycobacterial treatment.

Investigations Detection of rapid responders: Biomarkers, tissue mycolactone concentration and immune response will be measured at baseline. The rate of healing will be estimated by documenting the initial size of the lesion and the time to complete healing as previously (2).

Detection of Mu: Swabs homogenates will be inoculated onto Lowenstein Jensen slopes for culture and microscopy will be carried out on Ziehl-Neelsen stained smears for AFB. PCR for IS2404 will be carried out as described previously (3).

Biomarkers:

Serum samples will be subjected to multi-analyte profiling using Luminex multianalyte profiling to identify markers of oedematous disease, paradoxical reactions and rapid responders.

We will also use mass spectrometry-based proteomics to generate additional serum/tissue biomarkers taking a three-stage approach. First we will use sample fractionation and mass spectrometry (matrix-assisted laser desorption/ionisation/time of flight/mass spectrometry) to determine the degree of variability of proteomic composition in samples from subjects to be treated with antibiotics. This first screening will allow the identification and removal of subjects showing a partial response and subsequent analysis of those showing the most disparate responses. Stage 2 comprises a deep liquid chromatography mass spectrometry (LC/MS/MS)-based quantitative analysis of pooled samples (3 pools generated randomly from each response cohort) from each of the identified response groups. Molecules that show significant changes will be considered as candidate biomarkers of drug response. In Stage 3 immunoassays (ELISA) will be developed in order to test the validity of each novel biomarker in its ability separately or in combination with existing biomarkers to predict drug response.

Immune response: Whole blood samples will be incubated with Mu antigens overnight at 37 degrees celsius and the supernate will be stored for cytokine assays using ELISA as in our previous studies (4).

Antigen stimulated T cell populations will also be studied by flow cytometry to assess the proportion of Interferon(IFN) gamma, Tumor necrosis factor (TNF) and interleukin-2 (IL2) secreting T cells in patients compared to controls.

Mycolactone detection: Lipids will be extracted from homogenised skin biopsies and swabs//fine needle aspirates and the biological activity of mycolactone will be measured by a cytotoxicity assay as described previously using human embryonic lung fibroblasts as target cells. The presence of mycolactone in tissue samples will be confirmed and quantified by mass spectrometry as previously described (5). Mycolactone production by the strain of Mu isolated from oedematous lesions will be quantified in vitro and the tissue concentration of mycolactone in oedematous lesions will be measured.

Sample size and justification There will be 450 participants in this study. Our previous studies showed a mean difference in TNF alpha at baseline between fast and slow responders to be 15pg/ml and a standard deviation of 33pg/ml. The standardized mean difference computed as d=15/33 was 0.45. The sample size required to detect this difference with a two-sided significance of 5% and with 80% power would be 100 participants in each group (that 200 patients). We expect an attrition rate of 20% bringing the sample size to 250 patients. There will be control group of 200 healthy volunteers

Statistical analysis For the purpose of this study a "rapid responder or fast responder" is defined as a patient with a time to healing of less than 12 weeks or rate of healing of greater than 4mm/week and " slow responder or slow healer" is defined as a patient with time to healing of 12 or more weeks or rate of healing of less than 3 mm/week

Data generated by multianalyte profiling will be analyzed by multivariate analysis, including principal component analysis (PCA) and partial least-squares (PLS)-related methods, using the SIMCA 13 software (Umetrics, Sweden) . Univariate analyses will be performed to further characterize candidate biomarkers. Here, differences between controls and disease patients will be analyzed using the non-parametric Wilcoxon rank sum (Mann-Whitney) test. Paired samples for BUD patients at week 0 and week 12 will be compared using the Wilcoxon signed rank test. Univariate analysis and multiple testing adjustments will be performed using R software (version 2.13.2, R Development Core Team, R Foundation for Statistical Computing, Vienna, Austria) and package QVALUE. GraphPad Prism software will be used for graphical representation.

ELIGIBILITY:
Inclusion Criteria:

* All patients 5 years old or more diagnosed as having Buruli ulcer.
* Age-matched household contacts of patients that present with Buruli ulcer and healthy volunteers living in Buruli ulcer non-endemic communities

Exclusion Criteria:

* Patients aged less than 5 years and those
* Unwilling to give informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed Buruli ulcer and healthy contacts of patients with Buruli ulcer
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12-15 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum/plasma proteins in diseased and healthy subjects | Assessed for diseased participants at baseline, 8, 12, 16 weeks and only at baseline for healthy subjects

SECONDARY OUTCOMES:
Viable M. ulcerans and bacterial load measurement in tissue of diseased subjects | Assessed at baseline, 4, 8, 12, 16 only if lesions are not healed

OTHER OUTCOMES:
Mycolactone measurement in tissue of diseased subjects | Assessed at baseline, 4, 8, 12, 16 only if lesions are not healed
Rate of healing and time to healing in diseased subjects | The primary outcome measure will be assessed for each participant at the time of healing which will vary for participants

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Phillips, FWACP,FGCP, Principal Investigator — Kwame Nkrumah University of Science and Technology
Locations (3):
- Ghana (3):
  - Tepa Government Hospital, Tepa, Ahafo Ano North District
  - Agogo Presbyterian Hospital, Agogo, Asante Akim North District
  - Nkawie Government Hospital, Nkawie, Atwima Nwabiangya District

REFERENCES:
- [Derived] Frimpong M, Agbavor B, Duah MS, Loglo A, Sarpong FN, Boakye-Appiah J, Abass KM, Dongyele M, Amofa G, Tuah W, Frempong M, Amoako YA, Wansbrough-Jones M, Phillips RO. Paradoxical reactions in Buruli ulcer after initiation of antibiotic therapy: Relationship to bacterial load. PLoS Negl Trop Dis. 2019 Aug 26;13(8):e0007689. doi: 10.1371/journal.pntd.0007689. eCollection 2019 Aug. PMID 31449522